CLINICAL TRIAL: NCT01103986
Title: Assessing the Effectiveness of a Health Literacy Intervention in the Workplace: A Quasi-experimental Pre-post Randomized Controlled Study
Brief Title: Assessing the Effectiveness of a Health Literacy Intervention in the Workplace
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 0912-255X
Record Dates: First submitted 2010-02-01; First posted 2010-04-15 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Health Literacy
Keywords: health literacy; consumer health information; patient education as topics/methods; patient participation
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention)
- motivational/ health literacy education (Experimental)
  Interventions: Behavioral: Motivational/health literacy education (Test group)

INTERVENTIONS:
Behavioral: Motivational/health literacy education (Test group) — Attend a 1-hour class to learn how to use the book "What to Do When Your Child Gets Sick."
  Arms: motivational/ health literacy education

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a health literacy/motivational intervention in a workplace setting. Parents will be taught how to use a child health book to lessen inappropriate use of physician services and improve parent confidence in their ability to identify and obtain necessary assistance when their children are ill.

ELIGIBILITY:
Inclusion Criteria:

* currently employed at the Children's Mercy Hospitals and Clinics, MO or KS, or working under contract
* parent/legally authorized representative/primary care giver taking care of a child birth to 12 years old

Exclusion Criteria:

* non-English speaking and reading
* under 18 years old unless a minor parent
* a medical or nursing degree (MD, DO, Physician's Assistant, Nurse Practitioner, RN or LPN)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
number of non emergency room clinician visits | within 1 week prior to class and 90 days post-class
  Determine if parents/primary caregivers' attendance at a class to learn how to use a child health book leads to fewer non-emergency room clinician visits for their children.

SECONDARY OUTCOMES:
number of emergency department visits | within 1 week prior to class and 90 days post-class
  To determine if parents/primary caregivers attending a class to learn how to use a child health book leads to fewer emergency department visits
pre and post intervention measures of self-identified competency. | within 1 week prior to class and 90 days post-class
  To assess feelings of parents/primary caregiver competence in appropriately managing their children's illnesses using pre and post intervention measures of self-identified competency.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A Neilan, MT (ASCP), Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- The Children's Mercy Hospitals and Clinics, Kansas City, Missouri, United States

REFERENCES:
- [Background] Bryan C. Provider and policy response to reverse the consequences of low health literacy. J Healthc Manag. 2008 Jul-Aug;53(4):230-41. PMID 18720685
- [Background] Ensuring Positive Health Outcomes in Head Start Children and Famiies Pilot Study, Executive Summary. Herman A, September 2002